CLINICAL TRIAL: NCT04994366
Title: Increasing Patient Experience Survey Responses
Status: Completed | Type: Observational
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Other Study IDs: QI-NYUPatientExperience
Record Dates: First submitted 2021-07-30; First posted 2021-08-06 (Actual); Last update posted 2022-10-10 (Actual); Status verified 2022-10

CONDITIONS: Patient Satisfaction
MeSH Terms: conditions — Patient Satisfaction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Intervention Group: The cohort receiving Thank you cards during their stay.
  Interventions: Other: Thank you card
- Control Group: The cohort not receiving thank you cards during their stay.

INTERVENTIONS:
Other: Thank you card — A card thanking the patient for choosing NYU and entrusting us with their care. The card notifies the patient that they may receive a patient satisfaction survey after discharge.
  Groups: Intervention Group

SUMMARY:
This project aims to evaluate the effect of thank you cards on patient experience survey response rate.

ELIGIBILITY:
Inclusion Criteria:

* All patients who have been discharged from the designated hospital units during the study period

Exclusion Criteria:

* N/A

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients who have been discharged from the designated hospital units during the study period
Sampling Method: Probability Sample
Enrollment: 929 (Actual)
Dates: Start 2021-07-12 (Actual); Primary Completion 2021-11-14 (Actual); Study Completion 2021-11-14 (Actual)

PRIMARY OUTCOMES:
Survey response rate | 1 year
  The rate at which patients complete and submit the patient satisfaction survey

CONTACTS AND LOCATIONS:
Overall Officials: Leora Horwitz, MD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States